CLINICAL TRIAL: NCT04925609
Title: A Phase I/II Study of Brigatinib in Pediatric and Young Adult Patients With ALK+ Anaplastic Large Cell Lymphoma, Inflammatory Myofibroblastic Tumors or Other Solid Tumors
Brief Title: Brigatinib in Pediatric and Young Adult Patients With ALK+ ALCL, IMT or Other Solid Tumors
Acronym: Briga-PED
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Princess Maxima Center for Pediatric Oncology (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ITCC-098
Record Dates: First submitted 2021-05-17; First posted 2021-06-14 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-10

CONDITIONS: Anaplastic Large Cell Lymphoma, ALK-Positive; Inflammatory Myofibroblastic Tumor; Other Solid Tumor
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic; Granuloma, Plasma Cell | interventions — brigatinib

STUDY DESIGN:
Intervention Model Description: Phase 1:
  * To estimate the MTD/RP2D regimen of brigatinib monotherapy when administered in pediatric and AYA patients with ALK+ ALCL or ALK+ solid tumors.
  * To characterize the PK of brigatinib administered as monotherapy in pediatric and AYA patients with ALK+ ALCL or ALK+ solid tumors.
  Note that:
  * If the MTD is not reached at the highest proposed test dose, no further dose-escalation will be performed.
  * Pediatric PK data, compared to exposure in adults, and cumulative toxicity, will be taken into consideration to determine the RP2D regimen.
  Phase 2:
  • B1, ALK+ IMT: To establish the activity (ORR by RECIST 1.1) of single agent brigatinib when administered to children with ALK+ IMT.
  • B2, ALK+ ALCL: To establish the efficacy (EFS) of single agent brigatinib when administered to children with ALK+ ALCL for a duration of 2 years, without SCT in consolidation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1 (Other): Phase 1:
  * To estimate the MTD/RP2D regimen of brigatinib monotherapy when administered in pediatric and AYA patients with ALK+ ALCL or ALK+ solid tumors.
  * To characterize the PK of brigatinib administered as monotherapy in pediatric and AYA patients with ALK+ ALCL or ALK+ solid tumors.
  Note that:
  * If the MTD is not reached at the highest proposed test dose, no further dose-escalation will be performed.
  * Pediatric PK data, compared to exposure in adults, and cumulative toxicity, will be taken into consideration to determine the RP2D regimen.
  Interventions: Drug: Brigatinib
- Phase 2 (Other): Phase 2:
  • B1, ALK+ IMT: To establish the activity (ORR by RECIST 1.1) of single agent brigatinib when administered to children with ALK+ IMT.
  • B2, ALK+ ALCL: To establish the efficacy (EFS) of single agent brigatinib when administered to children with ALK+ ALCL for a duration of 2 years, without SCT in consolidation.
  Interventions: Drug: Brigatinib

INTERVENTIONS:
Drug: Brigatinib — Brigatinib is a second generation novel, orally administered, tyrosine kinase inhibitor (TKI) that potently inhibits activated variants of ALK and to a lesser extent ROS1.
  Other Names: Alunbrig

SUMMARY:
This is an open-label, phase I-II dose-escalation and expansion study designed to define the recommended dose of brigatinib as monotherapy in pediatric and young adult patients with ALK+ ALCL, IMT or other solid tumors and to evaluate the pharmacokinetics (PK), (long-term) safety, and efficacy of brigatinib in these children.

DETAILED DESCRIPTION:
This is an open-label, phase I-II dose-escalation and expansion study designed to define the recommended dose of brigatinib as monotherapy in pediatric and young adult patients with ALK+ ALCL, IMT or other solid tumors and to evaluate the pharmacokinetics (PK), (long-term) safety, and efficacy of brigatinib in these children.

Phase 1 part will be a dose escalation part using a rolling-6 design, aiming to accrue a minimum of 6 and a maximum of 18 evaluable patients in two dose-levels (and minus 1), at least 2/3 of included patients will be ≤18 years.

Phase 2 will be the tumor cohort expansion part of the study to further evaluate the safety, tolerability, and clinical activity/efficacy of brigatinib as monotherapy in two tumor-specific cohorts:

* Cohort B1: ALK+ IMT Planned sample size for Phase 2 is 12 patients with IMT. Patients who are included in the monotherapy Phase 1 IMT dose-escalation portion of the study will be included in the expansion cohort analysis if they receive the RP2D, and will count towards the total sample size of 12 patients.
* Cohort B2: ALK+ ALCL Planned sample size for Phase 2 is 22 patients with ALCL. Patients who are included in the monotherapy Phase 1 ALCL dose-escalation portion of the study will be included in the expansion cohort analysis if they receive the RP2D, and will count towards the total sample size of 22 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 1 and < 26 years of age at the time of enrollment, and able to swallow brigatinib tablets at the time of enrollment, with a minimum weight of 10 kg. Note: for phase 1 only patients ≤18 years old will be eligible, A liquid formulation for children with a weight lower than 10 kg or for those that cannot swallow tablets is in development.
2. Patients must have a confirmed diagnosis of cancer histologically at baseline. In patients where a repeat biopsy at relapse (or moment of refractory disease) is considered not feasible by the treating physician, archived material from diagnosis needs to be available for central review.
3. Patients are required to provide prior results showing an activating ALK aberration in the tumor per local laboratory results, and material needs to be available for central laboratory confirmation of ALK status. For ALK+ ALCL, detection of ALK with immunohistochemistry (IHC) is sufficient for inclusion, all others require molecular evidence of a ALK fusion gene or mutation by FISH, PCR or NGS. ALK detection will be confirmed centrally with FISH.
4. For Phase 1:

   * Patients with ALCL must be relapsed/refractory or intolerant to standard therapies. Refractory disease for ALCL is defined as:

     o no response to ALCL99/other standard of care chemotherapy (SD or PD of measurable lesions), and/or

     o MRD-positivity by qualitative PCR for NPM-ALK prophase after one block ALCL99/other standard of care chemotherapy (before the second course of chemotherapy).
   * Patients with relapsed/refractory (R/R) IMT must not be suitable for curative surgical resection without causing mutilation. Newly diagnosed patients with unresectable ALK+ IMT, or when surgery would imply severe mutilation may also be included, as well as metastatic disease.
   * Patients with other solid tumors (excluding IMT) must have relapsed or refractory disease.
5. For Phase 2, patients must have measurable and/or evaluable disease:

   * Patients with ALCL must be relapsed/refractory. Refractory disease for ALCL is defined as:

     * no response to ALCL99/other standard of care chemotherapy (SD or PD of measurable lesions), and/or
     * MRD-positivity by qualitative PCR for NPM-ALK prophase after one block ALCL99/other standard of care chemotherapy (before the second course of chemotherapy).
   * Patients with R/R IMT Relapsed/refractory ALK+ IMT, or newly diagnosed, including advanced and metastatic, ALK+ IMT which cannot be surgically resected without causing mutilation
6. Performance Status: Karnofsky performance status ≥40% for patients >16 years of age or Lansky Play Scale ≥40% for patients ≤16 years of age.
7. Patients must not be receiving other investigational medications (defined as medicinal products not yet approved for any indications, including alternative/herbal therapies) within 30 days of first dose of study drug or while on study.
8. For patients receiving prior therapy:

   * Patients who already received previous treatment with ALK inhibitors except for brigatinib can be included in this study.
   * Patients must have recovered to Grade <2 NCI CTCAE v5.0 or to baseline, from any nonhematologic toxicities (except alopecia and peripheral neuropathy) due to previous therapy.
   * Patients who relapsed while receiving cytotoxic therapy: at least 14 days must have passed since the completion of the last dose of chemotherapy before the first dose of brigatinib can be given.
   * Patients who have experienced relapse after a prior HSCT are eligible, provided they have no evidence of acute or chronic graft-versus-host disease (GVHD), are not receiving GVHD prophylaxis or treatment, and are at least 45 days posttransplant at the time of enrollment.
   * Hematopoietic growth factors: before the first dose of brigatinib, at least 7 days must have passed since completion of therapy with granulocyte colony-stimulating factor or other growth factors, and at least 14 days must have passed since completion of therapy with pegfilgrastim.
   * Biologics and Targeted Therapies:

     o Immunotherapy: Before the first dose of brigatinib, at least 30 days must have passed after the completion of any type of immunotherapy, (i.e. monoclonal antibodies [anti-PD1/PDL1], tumor vaccines, chimeric antigen receptor [CAR] T cells, etc.).

     o Other: before the first dose of brigatinib, at least 7 days must have passed since the last dose of a biologic agent. For agents that have known adverse events (AEs) occurring beyond 7 days after administration, this period must be extended beyond the time during which AEs are known to occur. The duration of this interval must be discussed with the sponsor's medical monitor/designee.

     o Immunosuppressive therapy: Before the first dose of brigatinib, at least 14 days must have passed after the completion of immunosuppressive therapy (including regimens following stem cell transplant).

     o For symptomatic patients that urgently need relief (i.e. airway obstruction), therapeutic doses of corticosteroids may be administered for a short course (up to 5 days).

     o Radiotherapy (XRT): No washout period is necessary for radiation given to any extramedullary site other than the CNS and lungs; ≥45 days must have passed if patient received prior total body irradiation or craniospinal or cranial XRT; ≥28 days must have passed if patient received radiotherapy to the lung. For patients receiving XRT to both lungs, or in case of stereotactic radiotherapy, the PIs should be consulted before inclusion.
9. Patients must meet the organ function and system function requirements as stated below:

   * Patients must have adequate renal and hepatic function as indicated by the following laboratory values:

     o Patient's serum creatinine must be ≤ 1.5 x institutional upper limit of normal (ULN) according to age. If the serum creatinine is greater than 1.5 x institutional ULN, the patient must have a radioisotope GFR ≥ 70mL/min/1.73m2
     * Adequate liver function defined as: direct bilirubin ≤1.5 times the upper limit of normal (ULN) for age AND AST and ALT must be ≤5 times the ULN for age (unless related to involvement of the liver or histiocytic/macrophage inflammatory process).
   * No clinical, radiological or laboratory evidence of pancreatitis, including o Serum lipase must be <2 × the ULN, and

     o Serum amylase must be <2 × the ULN.
   * Absolute neutrophil count: ≥0.75 × 10 9/L, except in case of macrophage activation syndrome (MAS) or bone marrow involvement.
   * Platelet count o In phase 1: Platelet count: ≥75 × 10^9/ L, except in case of MAS or bone marrow involvement o In phase 2: : Platelet count: ≥75 × 10^9/ L, except in case of MAS or bone marrow involvement. For patients post SCT, platelet count ≥50 × 10^9/ L is accepted.Hemoglobin ≥8 g/dL or 5.0 mmol/L (red blood cell [RBC] transfusions to achieve this value are allowed with the condition that the patient has no signs of active bleeding or hemolysis).
10. Adequate cardiac function defined as shortening fraction ≥27% by echocardiogram OR left ventricular ejection fraction of ≥50% by multigated acquisition scan.
11. Normal QT interval corrected per Fridericia method (QTcF) on screening electrocardiogram (ECG), defined as QTcF of ≤450 ms.
12. Have a life expectancy of ≥3 months.
13. Female patients of childbearing potential must have a negative urine or serum pregnancy test confirmed prior to enrollment.
14. Female patients with infants must agree not to breastfeed their infants while on this study.
15. Contraception:

    • Male and female patients of child-bearing potential must agree to use, an effective method for male and highly effective method for female, of contraception approved by the investigator during the study, following the CTFG recommendations, for at least 8 months for females and for at least 5 months for males after the last dose of brigatinib.

    • Highly effective methods of contraception include (but not exclusively) the following contraceptive methods:

    o combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation
    * progestogen-only hormonal contraception associated with inhibition of ovulation
    * intrauterine device (IUD), intrauterine hormone-releasing system (IUS), sexual abstinence.
16. Voluntary written informed consent according to law and regulations

    -

Exclusion Criteria:

Patients meeting any of the following exclusion criteria are not to be enrolled in the study:

1. Patients receiving systemic treatment with strong or moderate CYP3A inhibitors or inducers within 14 days or five half-life times whichever the less prior to the first dose of study drug (refer to Section 5.2 for a list of example medications).
2. Diagnosis of another concurrent primary malignancy.
3. Clinically significant cardiovascular disease, including any of the following:

   * Myocardial infarction or unstable angina within 6 months of study entry.
   * History of or presence of heart block, and/or clinically significant ventricular or atrial arrhythmias.
   * Uncontrolled hypertension defined as persistent elevation of systolic and/or diastolic blood pressures to ≥95th percentile based on age, sex, and height percentiles despite appropriate antihypertensive management.
4. Planned non-protocol chemotherapy, radiation therapy, another investigational agent, or immunotherapy while patient is on study treatment.
5. Any illness that affects gastrointestinal absorption.
6. Ongoing or active systemic infection, active seropositive HIV, or known active hepatitis B or C infection.
7. Any pre-existing condition or illness that, in the opinion of the investigator or sponsor, would compromise patient safety or interfere with the evaluation of the safety or efficacy of brigatinib.
8. Patients with a history of cerebrovascular ischemia/hemorrhage with residual deficits are not eligible (patients with a history of cerebrovascular ischemia/hemorrhage remain eligible provided all neurologic deficits have resolved).
9. Uncontrolled seizure disorder (patients with seizure disorders that do not require antiepileptic drugs, or are well controlled with stable doses of antiepileptic drugs are eligible).

Ages: 1 Year to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 65 (Estimated)
Dates: Start 2022-08-18 (Actual); Primary Completion 2033-12 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
Phase 1: assess the MTD/RP2D regimen | 2 years
  Phase 1:
  • To assess the MTD/RP2D regimen of brigatinib monotherapy when administered in pediatric and AYA patients with ALK+ ALCL or ALK+ solid tumors.
  Dose-limiting toxicities (DLTs) during the first course of therapy.
  The RP2D is defined as the dose that results in equivalent (approximately ±20% of the adult values) PK exposure to 180 mg QD with a 7 day lead in of 90 mg QD in adults and with 0 or 1 DLT in 6 patients.
Phase 1: to characterize the PK of brigatinib | 2 years
  Phase 1:
  • To characterize the PK of brigatinib administered as monotherapy in pediatric and AYA patients with ALK+ ALCL or ALK+ solid tumors:
  o maximum observed concentration (Cmax),
Phase 1: to characterize the PK of brigatinib | 2 years
  Phase 1:
  • To characterize the PK of brigatinib administered as monotherapy in pediatric and AYA patients with ALK+ ALCL or ALK+ solid tumors:
  o area under the concentration-time curve from time 0 to the time of the last quantifiable concentration (AUClast).
Phase 1: to characterize the PK of brigatinib | 2 years
  Phase 1:
  * To characterize the PK of brigatinib administered as monotherapy in pediatric and AYA patients with ALK+ ALCL or ALK+ solid tumors:
    * time of first occurrence of maximum observed concentration (Tmax), T ½.
Phase 2: ORR in IMT | 2 years
  • B1, ALK+ IMT:
  To establish the activity (ORR by RECIST 1.1, best response) of single agent brigatinib when administered to children with ALK+ IMT:
  Best response, defined as the percentage of patients with CR or PR according to RECIST 1.1 as best response during brigatinib treatment.
Phase 2: EFS in ALCL | 2 years
  • B2, ALK+ ALCL: To establish the efficacy (EFS) of single agent brigatinib when administered to children with ALK+ ALCL for a duration of 2 years, without SCT in consolidation.
  EFS, defined as the time between start of study treatment and first event being progressive disease (according to IPNHL criteria), relapse, death of any cause and second malignancies.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Zwaan, Prof, Principal Investigator — Princess Maxima Center for Pediatric Oncology in The Netherlands
Locations (2):
- Institut Gustave Roussy, Paris, France
- Princess Máxima Center for Pediatric Oncology, Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: CSR
Time Frame: The CSR will be made available within 6 months upon study end.
Access Criteria: A summary of the study results will be made public via clinicaltrials.gov as well as to Ethical committees/ Health Authorities and all participating patients by providing them through their treating physicians a patient letter with a summary of the results.